CLINICAL TRIAL: NCT06653400
Title: Combined Ketorolac and Lidocaine Paracervical Block for Office Hysteroscopy: a Randomized Controlled Trial
Brief Title: Combined Ketorolac and Lidocaine Paracervical Block for Office Hysteroscopy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Charles Ascher-Walsh, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY-23-01631
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-09

CONDITIONS: Abnormal Uterine Bleeding; Analgesia; Paracervical Block
MeSH Terms: conditions — Metrorrhagia; Agnosia | interventions — Anesthesia, Obstetrical; Lidocaine; Ketorolac

STUDY DESIGN:
Intervention Model Description: To study the effect of a combined ketorolac and lidocaine paracervical block on procedure related pain with office hysteroscopy. The standard of care is currently just a lidocaine paracervical block.
Who Masked: Participant, Care Provider
Masking Description: An assistant will be in charge of mixing either the intervention or control paracervical block. The physician performing the procedure and the patient will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lidocaine alone (Placebo Comparator): Paracervical block will be performed with just lidocaine
  Interventions: Procedure: paracervical block; Drug: Lidocaine
- Lidocaine plus ketorolac (Experimental): Paracervical block will be performed with lidocaine plus ketorolac
  Interventions: Procedure: paracervical block; Drug: Lidocaine; Drug: ketorolac

INTERVENTIONS:
Procedure: paracervical block — paracervical block with office hysteroscopy
Drug: Lidocaine — Dosage: 20 mL of 1% lidocaine
Drug: ketorolac — Dosage: 2 mL (30 mg) of ketorolac
  Arms: Lidocaine plus ketorolac

SUMMARY:
A randomized double-blind placebo controlled trial comparing the effect of a combined ketorolac and lidocaine paracervical block with a standard lidocaine paracervical block on procedure related pain with office hysteroscopies.

DETAILED DESCRIPTION:
A randomized double-blind placebo controlled trial comparing the effect of a combined ketorolac and lidocaine paracervical block with a standard lidocaine paracervical block on procedure related pain with office hysteroscopies. Primary Objective: To study the effect of a combined ketorolac and lidocaine paracervical block on procedure related pain with office hysteroscopy. Secondary Objectives: To study the effect of a combined ketorolac and lidocaine paracervical block on patient satisfaction and post procedure pain. To assess for major adverse events with the use of a combined ketorolac and lidocaine paracervical block for office hysteroscopy when compared with a standard lidocaine paracervical block. Primary Endpoint: Pain on a 100 mm visual analogue scale during cervical dilation. Secondary Endpoints: Pain on a 100 mm visual analogue scale during the paracervical block, during the office hysteroscopy, immediately after the hysteroscopy, and 30 minutes after the procedure. Other secondary endpoints include patient satisfaction, frequency of procedure termination, and adverse events. Patients assigned female at birth, booked for office hysteroscopy at Mount Sinai Hospital faculty practice associates. Patients scheduled for office hysteroscopy through seeing a Gynecologist at either 5 E 98th Street Faculty Practice Associates or 1176 5th Avenue Gynecology Practice. 5 E 98th Street primarily cares for privately insured patients, while 1176 5th Avenue cares for a mix of privately insured as well as patients insured with Medicaid. Regardless of recruitment site, all office hysteroscopies will be performed at the 5 E 98th Street facility. A randomized controlled trial designed to investigate if ketorolac added to a paracervical block reduces procedure related pain. Patient will be randomized to a standard paracervical block versus a paracervical block with ketorolac added. The study will be conducted over two years. Patients will be followed for the duration of the two-year study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients assigned female at birth,
* booked for office hysteroscopy at Mount Sinai Hospital faculty practice associates.

Exclusion Criteria:

* Allergy to ketorolac or non-steroidal anti-inflammatory medications
* Allergy to lidocaine
* Presence of thrombocytopenia
* Contraindications to lidocaine
* History of gastritis or gastric ulcer
* Acute renal failure or chronic renal disease
* Chronic liver disease
* History of bleeding diathesis
* Long term narcotic use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain visual analogue scale (VAS) | during procedure (cervical dilation)
  Pain as measured on a 100 mm visual analogue scale (VAS) with cervical dilation.
  Full scale scored from 0-100, higher score indicates more pain.

SECONDARY OUTCOMES:
Pain visual analogue scale (VAS) | with paracervical block, during procedure, immediately after procedure, thirty minutes after the procedure
  Pain as measured on a 100 mm visual analogue scale (VAS). Full scale scored from 0-100, higher score indicates more pain..
Patient Satisfaction | with paracervical block, during procedure, immediately after procedure, thirty minutes after the procedure
  Full scale scored from 0-100, higher score indicates (better or poorer) health outcomes.
Frequency of procedure termination | with paracervical block, during procedure, immediately after procedure, thirty minutes after the procedure
  Number of times of procedure termination

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ascher-Walsh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data. To achieve aims in the approved proposal. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.